CLINICAL TRIAL: NCT06198426
Title: A Phase 1/2, Multicenter, Open-label Study of IBI3004 in Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of IBI3004 in Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The company's development strategy has been adjusted
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI3004A101
Record Dates: First submitted 2023-12-24; First posted 2024-01-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI3004 (Experimental)
  Interventions: Drug: IBI3004

INTERVENTIONS:
Drug: IBI3004 — IBI3004 will be administered. The Dose Limiting Toxicity (DLT) will be observed in the first treatment cycle. After completion of the DLT observation period, subjects will continue to receive IBI3004 until death, disease progression, intolerable toxicity, start of a new anticancer treatment, withdrawal of consent for study participation, end of the study, or for a maximum of 24 months, whichever occurs first.

SUMMARY:
This is an open-label, multicenter, dose escalation and expansion phase I /II study of IBI3004 in subjects with unresectable, locally advanced or metastatic solid tumors. It includes a phase 1 dose escalation and expansion section to identify Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of IBI3004. Accelerated titration and the Bayesian Optimal Interval (BOIN) design is used to find the MTD or RP2D, and the maximum sample size is 46. One or more dose levels will be selected for dose expansion, each dose group will be expanded to 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. Male or female subjects ≥ 18 years old. For Part 1, age ≥18 and ≤75 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
4. Anticipated life expectancy of ≥ 12 weeks;
5. Adequate bone marrow and organ function

Exclusion Criteria:

1. Enrolled in any other interventional clinical research except unless only involved in an observational study (non-interventional) or in the follow-up phase of an interventional study;
2. Received previous anti-tumor therapy: within 21 days of monoclonal antibodies or cytotoxic therapy prior to the first dose of the study drug, or within 14 days of small molecule targeted drugs prior to the first dose of the study drug. Received palliative radiation therapy within 2 weeks prior to the first dose of the study drug, or received radical radiation therapy within 4 weeks prior to the first dose of the study drug;
3. Received live vaccines within 4 weeks prior to first administration of the study drug or plan on receiving any live vaccine during the study;
4. Has adverse reactions resulting from previous antitumor therapies, which have not resolved to Grade 0 or 1 toxicity according to NCI-Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (except for alopecia, fatigue, pigmentation and other conditions with no safety risk according to investigator' discretion) or baseline prior to the first dose of the study drug;
5. Undergone major surgery (Craniotomy, thoracotomy or laparotomy, and other surgery according to investigator' discretion, excluding needle biopsy) within 4 weeks prior to the first dose of the study drug, or who are expected to undergo major surgery during the study period, or who have severe unhealed wounds, trauma, ulcers, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 30 days post last dose
  Number of patients who experienced AEs from the first dose until 30 days after the last dose

SECONDARY OUTCOMES:
Dose limiting toxicities (DLTs) | Up to 28 days post first dose
  To evaluate the safety and tolerability of IBI3004

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (3):
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
- China (2):
  - Jiang Su Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No